CLINICAL TRIAL: NCT01077492
Title: CT-PET Virtual Bronchoscopy Guided Transbronchial Needle Aspiration for Mediastinal Lymph Node Staging in Suspected Lung Cancer
Brief Title: Virtual Bronchoscopy Transbronchial Needle Aspiration(TBNA): a Proof of Concept Study
Status: Terminated | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: T.G. Sutedja, MD, PhD, VU University Medical Center
Other Study IDs: 09/327
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2010-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; mediastinal lymph nodes; TBNA; staging lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected mediastianl lymph nodes: Patients with (suspected) lung cancer requiring MLN staging after CT-PET during routine work-up according to existing staging guidelines.
  Interventions: Other: Virtual Bronchoscopy Navigation

INTERVENTIONS:
Other: Virtual Bronchoscopy Navigation — Use of dedicated virtual bronchoscopy navigation software using 4D CT-PET scan spacial data.

SUMMARY:
The purpose of this study is to determine wether CT-PET virtual bronchoscopy guided transbronchial needle aspiration is suitable for the investigation of mediastinal lymph nodes which is needed for correct staging of lung cancer.

DETAILED DESCRIPTION:
Accurate staging of mediastinal lymph nodes (MLNs) in patients with lung carcinoma (LC) is paramount as the N stage largely determines treatment strategy, prognosis and outcome. Surgical staging such as mediastinoscopy is considered the gold standard. A less invasive alternative is transbronchial needle aspiration (TBNA). This technique is limited however by moderate and operator dependent accuracy. Recently less invasive strategies such as esophageal ultrasound guided fine needle aspiration (EUS-FNA) and endobronchial ultrasound guided TBNA (EBUS-TBNA) were introduced. These strategies have largely complemented TBNA and surgical staging, with high accuracy and low morbidity. Disadvantages compared to TBNA however are required specific expertise, higher equipment and maintenance costs, the need for more assisting personnel and the need for sedation. Advances in computer generated image processing based on available CT and PET images enable (quasi) real-time virtual bronchoscopy that can assist minimal invasive surgical performance including bronchoscopy. Optimizing the traditional TBNA procedure with these modern imaging techniques might be equally accurate and more cost effective.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Proven or suspected lung cancer, base on clinical picture and/or CT-PET findings
* Suspected involvement of mediastinal lymph nodes on CT-PET scan
* Written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected lung cancer requiring mediastinal lymph node staging after CT-PET scan during routine work-up according to local guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of VB in determining N2/N3 mediastinal lymph nodes | 1 year
  Feasibility of virtual bronchoscopy in showing the presence or abscense of N2/N3 mediastinal lymph node (MLN) metastasis with accuracy of 0.6 in puncturing MLN > 15 mm (CT images) and accuracy of 0.8 for MLN < 15 mm in the second phase of the study.

SECONDARY OUTCOMES:
Duration of the session within the optimal time window of local anesthesia using lidocaine 1%; comparable to standard routine bronchoscopic procedure on an outpatient basis, i.e. not exceeding 30 minutes. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Hashemi, MD, Study Chair — Amsterdam UMC, location VUmc; Hans Daniels, MD, Study Chair — Amsterdam UMC, location VUmc; Emiel Comans, PhD, Study Chair — Amsterdam UMC, location VUmc; Otto Hoekstra, PhD, Study Chair — Amsterdam UMC, location VUmc; Piet Postmus, PhD, Study Chair — Amsterdam UMC, location VUmc; Tom Sutedja, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands